CLINICAL TRIAL: NCT01398787
Title: Cosmetic Validation (US): AIR OPTIX® COLORS Among Habitual Wearers of FRESHLOOK®
Brief Title: Evaluation of the Cosmetic Performance of AIR OPTIX® COLORS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: P-383-C-004
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Cosmetic Appearance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIR OPTIX® COLORS (Experimental): Lotrafilcon B contact lens with color randomly assigned to one eye, with phemfilcon A contact lens with color in the fellow eye for contralateral wear
  Interventions: Device: Lotrafilcon B contact lens with color
- FRESHLOOK® COLORBLENDS (Active Comparator): Phemfilcon A contact lens with color randomly assigned to one eye, with lotrafilcon B contact lens with color in the fellow eye for contralateral wear
  Interventions: Device: Phemfilcon A contact lens with color

INTERVENTIONS:
Device: Lotrafilcon B contact lens with color — Plano (-0.00 diopter) silicone hydrogel contact lens in 1 of 4 colors: gray, blue, green, pure hazel
  Other Names: AIR OPTIX® COLORS
  Arms: AIR OPTIX® COLORS
Device: Phemfilcon A contact lens with color — Plano (-0.00 diopter) hydrogel contact lens in 1 of 4 colors: ColorBlends gray, Colorblends blue, Colorblends green, Colorblends pure hazel
  Other Names: FRESHLOOK® COLORBLENDS
  Arms: FRESHLOOK® COLORBLENDS

SUMMARY:
The purpose of this study was to evaluate the cosmetic performance of AIR OPTIX® COLORS contact lenses compared to FRESHLOOK® COLORBLENDS contact lenses in habitual FRESHLOOK® COLORBLENDS contact lens wearers.

DETAILED DESCRIPTION:
In this non-dispensing trial, each participant wore 4 pairs of color contact lenses (gray, blue, green, hazel) sequentially for less than 10 minutes each in a contralateral fashion (test lens in one eye, control lens in the other eye). Randomization took place for each of the 4 pairs of lenses as to which eye (left or right) wore the test and which wore the control. Participants were selected based on eye color (dark vs light/medium). The primary analysis population (AP1) was pre-specified as participants of any eye color who habitually wore FRESHLOOK® COLORBLENDS lenses in one of the four colors tested in this trial. Pair 1 lenses were dispensed per the participant's habitual lens color.

ELIGIBILITY:
Inclusion Criteria:

* Sign written Informed Consent document. If under legal age of consent, legally authorized representative must sign Informed Consent document and subject must sign Assent document.
* Have spectacles that provide acceptable near vision to wear over study lenses as needed to evaluate cosmetics of the lenses.
* Habitually wear FRESHLOOK® COLORBLENDS lenses at least two days per week.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks of enrollment in this trial.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Currently enrolled in any clinical trial.
* Evidence of systematic or ocular abnormality, infection, or disease which is likely to affect successful wear of contact lenses or use of accessory solutions as determined by the investigator.
* Any use of medications for which contact lens wear could be contraindicated as determined by the investigator.
* Other protocol-defined exclusion criteria may apply.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Holden Thomas, O.D., Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 18 US study centers.
Pre-assignment Details: Of the 198 enrolled participants, 1 was exited as a screen failure prior to study product exposure. This reporting group includes all enrolled and exposed participants (197).
Groups:
- AIR OPTIX® COLORS/FRESHLOOK® COLORBLENDS: AIR OPTIX® COLORS and FRESHLOOK® COLORBLENDS, contralateral wear
Period: Overall Study
Arm/Group | AIR OPTIX® COLORS/FRESHLOOK® COLORBLENDS
Started | 198
Completed | 197
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: The analysis population includes all enrolled and exposed participants.
Arm/Group | AIR OPTIX® COLORS/FRESHLOOK® COLORBLENDS
Number analyzed (Participants) | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Overall Preference
Description: The participant compared Pair 1 study lenses on eye and indicated overall preference using a 4-point Likert scale (prefer lens in the left eye, prefer lens in the right eye, no preference, or both eyes are equal). Overall preference is reported as the percentage of participants who preferred the study lens. Each lens was assessed separately. This outcome measure was pre-specified for Analysis Population 1 (AP1).
Time Frame: Day 1, 2-10 minutes after lens insertion
Population: The analysis population includes all enrolled and exposed participants in AP1, minus any discontinuations, missing responses, or protocol violations as determined by masked review.
Measure: Number; unit: Percentage of participants
Groups:
- AIR OPTIX® COLORS: Lotrafilcon B silicone hydrogel contact lens in 1 of 4 colors (gray, blue, green, pure hazel) worn in one eye for up to 10 minutes
- FRESHLOOK® COLORBLENDS: Phemfilcon A hydrogel contact lens in 1 of 4 colors (ColorBlends gray, Colorblends blue, Colorblends green, Colorblends pure hazel) worn in one eye for up to 10 minutes
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS
Number analyzed (Participants) | 168 | 168
Percentage of participants | 49.1 | 24.6

2. Primary Outcome: Initial Comfort Preference
Description: The participant compared the initial comfort (way it feels) of Pair 1 study lenses and indicated preference using a 4-point Likert scale (prefer lens in the left eye, prefer lens in the right eye, no preference, or both eyes are equal). Initial comfort preference is reported as the percentage of participants who preferred the study lens. Each lens was assessed separately. This outcome measure was pre-specified for Analysis Population 1 (AP1).
Time Frame: Day 1, 2 minutes after lens insertion
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS
Number analyzed (Participants) | 168 | 168
Percentage of participants | 55.1 | 23.4

3. Primary Outcome: Appearance Preference
Description: The participant compared the appearance (way it looks) of Pair 1 study lenses on eye and indicated preference using a 4-point Likert scale (prefer lens in the left eye, prefer lens in the right eye, no preference, or both eyes are equal). Appearance preference is reported as the percentage of participants who preferred the study lens. Each lens was assessed separately. This outcome measure was pre-specified for Analysis Population 1 (AP1).
Time Frame: Day 1, 2-10 minutes after lens insertion
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS
Number analyzed (Participants) | 168 | 168
Percentage of participants | 36.5 | 23.4

4. Primary Outcome: Subjective Rating of Initial Comfort
Description: The participant compared the initial comfort (way it feels) of Pair 1 study lenses and rated initial comfort using a 10-point scale (1=poor, 10=excellent). Each lens was assessed separately. This outcome measure was pre-specified for Analysis Population 1 (AP1).
Time Frame: Day 1, 2 minutes after lens insertion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS
Number analyzed (Participants) | 168 | 168
Units on a scale | 8.6 (1.9) | 7.5 (2.5)

5. Primary Outcome: Percent Positive Responses: Cosmetic Appearance (Strongly Agree, Agree)
Description: The participant compared the cosmetic appearance of Pair 1 study lenses on eye and answered 9 appearance-related questions using a 4-point Likert scale (strongly agree, agree, disagree, strongly disagree). The combined percentage of the top two responses (strongly agree, agree) is reported for each question. Each lens was assessed separately. This outcome measure was pre-specified for Analysis Population 1 (AP1).
Time Frame: Day 1, 2-10 minutes after lens insertion
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS
Number analyzed (Participants) | 168 | 168
Percentage of participants
  The lens looks natural on my eye | 84.9 | 77.0
  The lens makes my eye look bold | 78.9 | 81.3
  The lens makes my eye look bright | 81.3 | 75.8
  The lens makes my eye look beautiful | 89.1 | 84.9
  The lens makes my eye noticeable | 93.9 | 94.0
  The lens enhances my eye color | 81.9 | 78.8
  I like the way my eye looks | 89.1 | 84.8
  The lens makes me look beautiful | 84.9 | 83.1
  The lens transforms the color of my eye | 88.6 | 93.4

6. Primary Outcome: Percent Positive Purchase Intent (Definitely Would Buy, Probably Would Buy)
Description: The participant compared Pair 1 study lenses and indicated purchase intent by answering the following question, "Assuming these lenses were at a price you would expect to pay, how likely would you be to purchase these lenses?" using a 5-point Likert scale (definitely would buy, probably would buy, might or might not buy, probably would not buy, definitely would not buy). The combined percentage of the top two responses (definitely would buy, probably would buy) is reported. Each lens was assessed separately. This outcome measure was pre-specified for Analysis Population 1 (AP1).
Time Frame: Day 1, 2-10 minutes after lens insertion
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS
Number analyzed (Participants) | 168 | 168
Percentage of participants | 80.2 | 59.9

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (5 months). An AE was defined as any untoward device experience with investigational or marketed product, whether it was considered to be device related or not.
Description: The analysis population includes all enrolled and exposed participants.
Groups:
- AIR OPTIX® COLORS: Lotrafilcon B silicone hydrogel contact lens in 4 colors (gray, blue, green, pure hazel) worn in one eye, up to 10 minutes each
- FRESHLOOK® COLORBLENDS: Phemfilcon A hydrogel contact lens in 4 colors (ColorBlends gray, Colorblends blue, Colorblends green, Colorblends pure hazel) worn in one eye, up to 10 minutes each
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS
Serious Adverse Events (participants affected / at risk) | 0/197 | 0/197
Other Adverse Events (participants affected / at risk) | 0/197 | 0/197

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.